CLINICAL TRIAL: NCT02825966
Title: Heart Sounds Measurement Using the Wearable Cardioverter Defibrillator (HS-WCD): Study Protocol
Brief Title: Heart Sounds Measurement Using the Wearable Cardioverter Defibrillator (HS-WCD) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 90D0153
Record Dates: First submitted 2016-06-28; First posted 2016-07-07 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Each subject first wears the AUDICOR-AM device for 15 minutes while sitting. Then the AUDICOR device is removed and the subject wears the WCD for 12-16 hours. After the WCD wear period, the WCD device is removed and the subject wears the AUDICOR device again for 15 minutes.
Oversight: Data Monitoring Committee: No

ARMS (1):
- AUDICOR then LifeVest then AUDICOR (Other): First, assigned to wear AUDICOR device for 15 minutes. Then assigned to wear the WCD, including 6 hours of overnight wear. Total anticipated wear time with WCD is 12-16 hours. Finally, assigned to wear the AUDICOR device for another 15 minutes after finishing the WCD wear.
  Interventions: Device: AUDICOR then LifeVest then AUDICOR

INTERVENTIONS:
Device: AUDICOR then LifeVest then AUDICOR — Wearable Cardioverter Defibrillator to record acoustic cardiograph signals.

SUMMARY:
A prospective, validation study to evaluate the data accuracy of heart sounds recorded by the LifeVest® Wearable Cardioverter Defibrillator (WCD). These data will be compared with the heart sounds data recorded by an FDA-cleared device AUDICOR AM device.

DETAILED DESCRIPTION:
To conduct a prospective, validation study to evaluate the data accuracy of heart sounds recorded by the LifeVest® Wearable Cardioverter Defibrillator (WCD). To show equivalence, these data will be compared with the heart sounds data recorded by an FDA-cleared AUDCIOR AM device .

The study will enroll a minimum of 27 and a maximum of 35 subjects.

Participants will be adult patients (age ≥ 18 years) with at least seven patients over the age of 40 years. In addition, at least five patients with a history of heart failure will be included.

First, participants will wear the AUDICOR-AM device for 15 minutes while sitting quietly. Then, the AUDICOR device will be removed and the participants will wear the WCD for 15 minutes while sitting quietly. Next, while wearing the WCD, participants will perform various activities of daily living, including at least 6 hours of overnight wear. Finally, the WCD will be removed and the participants will wear the AUDICOR again for 15 minutes while sitting quietly.

This is a single center, prospective, observational study. This is a non-significant risk device study as all biological study parameters will be measured noninvasively with the WCD defibrillation capability disabled. In addition, the study device will not be used as a replacement for regularly prescribed therapies or diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers who are able to fit in the WCD garment (26 to 56 inches measured circumferentially at the level of the xiphoid process).
* Included in this group are at least five healthy subjects with a self-reported history of heart failure.
* The subject must be 18 years of age or older on the day of screening, with at least 7 subjects 40 years of age or older on the day of screening.

Exclusion Criteria:

* Mental, visual, physical, literacy, and auditory limitations that prevent interaction with the WCD equipment.
* Any acute medical conditions that prevent the following maneuvers: lying on back, lying on the right and left side, standing, sitting, and/ or leaning forward when sitting.
* Any self-reported shortness of breath, fatigue, swelling of feet, ankles, or legs, and/or chest pain
* Employees or family members of the sponsor.
* Unable or unwilling to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Szymkiewicz, MD, Study Director — VP Medical Affairs
Locations (1):
- MedPace Phase 1 Clinic, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AUDICOR AM Device, Then LifeVest, Then AUDICOR AM Device: First assigned to wear the AUDICOR device for 15 minutes. Then, assigned to wear the WCD during activities of daily living, including at least 6 hours of overnight wear. Total anticipated wear time with WCD is 12-16 hours. Finally, assigned to wear AUDICOR device for 15 minutes after finishing the WCD wear.
Period: Overall Study
Arm/Group | AUDICOR AM Device, Then LifeVest, Then AUDICOR AM Device
Started (Same 35 subjects wore the AUDICOR Ambulatory Monitoring (AM) and WCD devices sequentially.) | 35
Completed (Same 35 subjects wore the AUDICOR AM and WCD devices sequentially.) | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: First, all subjects are assigned to wear AUDICOR device for 15 minutes. Then they were assigned to wear the WCD, including 6 hours of overnight wear. Total anticipated wear time with WCD is 12-16 hours. Finally, they were assigned to wear the AUDICOR device for another 15 minutes after finishing the WCD wear.
Groups:
- AUDICOR AM Device, Then LifeVest, Then AUDICOR AM Device: Assigned to wear the AUDICOR device first, then the WCD, and finally the AUDICOR device again.
Arm/Group | AUDICOR AM Device, Then LifeVest, Then AUDICOR AM Device
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 35
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: To Establish Equivalence Between the Heart Sounds Data Recorded by the LifeVest and FDA-cleared AUDICOR AM System.
Description: Equivalence of the LifeVest device to the AUDICOR device was established by comparing the electromechanical activation time (EMAT) data of each device, collected during quiet sitting. The outcome was reported as the difference in EMAT measured by the LifeVest and AUDICOR device.
Time Frame: 15 minutes of sitting for each group of measurements (Audicor device, then LifeVest, then Audicor device again).
Population: All subjects participating in the study were adult patients (age ≥ 18 years).
Measure: Mean (Standard Deviation); unit: ms
Groups:
- AUDICOR AM Device (First) Wear: First, assigned to wear AUDICOR device for 15 minutes.
- LifeVest Wear: Subjects removed the AUDICOR device and wore the LifeVest device for 12-16 hours
- AUDICOR AM Device (Second) Wear: Subjects removed the LifeVest and then wore the AUDICOR AM device for 15 minutes
Arm/Group | AUDICOR AM Device (First) Wear | LifeVest Wear | AUDICOR AM Device (Second) Wear
Number analyzed (Participants) | 35 | 35 | 35
ms | 95.88 (17.5) | 96.98 (15.04) | 98.25 (19.11)
Statistical Analysis 1: Comparison: AUDICOR AM Device (First) Wear vs LifeVest Wear; First, the difference in EMAT between the LifeVest and AUDICOR device (first wear) was calculated for each subject. Then the mean and standard deviation of the differences in EMAT were calculated. The 2 devices were considered equivalent if the 90% confidence interval for mean difference in EMAT was within the pre-specified margin of [-12, 12] ms; Test type: Equivalence — The two one-sided t-test (TOST) was used to test equivalence. Using TOST, equivalence was established at α = 0.05 significance level if a (1-2α)*100% confidence interval for the average difference in EMAT (WCD-AUDICOR) was contained within the interval [-12, 12]; p < 0.001, two one-sided test (TOST); Mean Difference (Final Values) = 1.01, 90% CI 2-sided [-2.89 to 4.69]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a time period of 16 hours during which the testing with the LifeVest and the AUDICOR AM devices were performed. For the AUDICOR AM device, this includes the 15 minutes of use before the LifeVest was applied, as well as the 15 minutes of use after the LifeVest was removed (about 30 minutes total). For the LifeVest, this was about 15 to 16 hours of use.
Description: Because each subject wore both devices, adverse events are grouped by device (AUDICOR AM and LifeVest).
Groups:
- AUDICOR AM Device: All study subjects during the time the AUDICOR AM device was used.
- LifeVest: All study subjects during the time the LifeVest device was used.
Arm/Group | AUDICOR AM Device | LifeVest
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT02825966/Prot_SAP_000.pdf